CLINICAL TRIAL: NCT05244720
Title: Evaluation of Liver Disease in Individuals Attending Alcohol Abuse Treatment - a Randomized Controlled Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SJ-934
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2022-01

CONDITIONS: Liver Diseases
Keywords: alcohol; pilot study; feasibility
MeSH Terms: conditions — Liver Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Pilot study to determine feasibility
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Baseline questionnaire filled out at recruitment. Invited to an examination of the liver, by fibroscan and blood samples, shortly after recruitment.
  Follow-up by phone after 6 months.
  Interventions: Diagnostic Test: Fibroscan; Diagnostic Test: Blood samples
- Control (Other): Baseline questionnaire filled out at recruitment. Follow-up by phone after 6 months. Invited to an optional examination of the liver, by fibroscan and blood samples, after 6 months.
  Interventions: Diagnostic Test: Fibroscan; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Fibroscan — A percutaneous scan, that measures shear wave velocity. It estimates liver stiffness.
  Other Names: Transient elastography
Diagnostic Test: Blood samples — Blood samples to asses the function of liver, kidney and bone marrow, as well as nutrition/vitamin status.

SUMMARY:
This pilot study aims to evaluate the feasibility of a non-blinded randomized controlled trial with a parallel group design of an invitation to an evaluation of liver disease (intervention) compared to standard care with no invitation, among individuals in alcohol abuse treatment.

DETAILED DESCRIPTION:
Alcohol-related liver disease (ALD) is responsible for about 80% of all liver disease in Denmark. The prognosis for ALD is good, if detected early and abstinence is obtained. Unfortunately ALD is often diagnosed at a late state and the 1-year survival is only 30%.

Currently there is no available systematic screening for fibrosis/cirrhosis among patients with longterm abuse of alcohol and thereby high risk for developing ALD.

Transient elastography (TE) is a non-invasive, risk free and quick method of detecting fibrosis. TE is validated for diagnosing fibrosis and ruling out cirrhosis.

40 patients will be enrolled in the study with a 1:1 randomization. Baseline data is collected and informed concent is obtained at the local alcohol abuse treatment center, Novavi Køge. The fibroscan and blood samples are done at Zealand University Hospital, Køge. Follow-up is done after 6 months, by a project nurse, blinded to the intervention.

If the study proves to be feasible, our aim is to extend the study in order to investigate wether the interventions described above, could help decrease alcohol consumption/maintain abstinence for patients in alcohol treatment. Moreover the prevalence of fibrosis and cirrhosis found by fibroscan is examined.

ELIGIBILITY:
Inclusion Criteria:

* must be enrolled at alcohol treatment center Novavi Koege, Denmark
* Maximum 6 months of treatment at Novavi Koege

Exclusion Criteria:

* known severe liver disease
* life expectancy less than 6 months
* unable to give informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  >50% of those invited to participate gives written consent.
Retention | 6 months
  >50% of those recruited and randomized to an examination, will attend for an examination at the hospital
Completion | 6 months after randomization
  >50% of randomized patients complete follow-up

SECONDARY OUTCOMES:
Reduction in Number of heavy drinking days | 10 months
  Reduction in Number of heavy drinking days, data collected at follow-up after 6 months, compared to baseline data.
Abstinence or reduction in alcohol consumption | 10 months
  Abstinence from alcohol in the three months prior to the 6-months follow-up phone call.
Prevalence of fibrosis/cirrhosis in individuals in alcohol treatment | 6 months
  Results from fibroscan, with a mean value of >8 indicating fibrosis and a mean value of >15 indicating cirrhosis.
Reduction in AUDIT score | 10 months
  AUDIT score is reported at baseline, and again at the 6 months follow up phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Gro Askgaard, PhD, Study Chair — Department of Medicine, Zealand University Hospital; Lone Madsen, PhD, Principal Investigator — Department of Medicine, Zealand University Hospital
Locations (1):
- Department of Medicine, Zealand University Hospital, Køge, Denmark

REFERENCES:
- [Derived] Jepsen P, von Wowern N, Madsen LG, Klausen MK, During S, Benthien KS, Winther-Jensen M, Petersen J, Askgaard G. The LIVER CARE trial - screening for liver disease in individuals attending treatment for alcohol use disorder: a randomized controlled feasibility trial. Pilot Feasibility Stud. 2024 May 16;10(1):78. doi: 10.1186/s40814-024-01504-5. PMID 38755732